CLINICAL TRIAL: NCT04336410
Title: Phase 1 Open-label Study to Evaluate the Safety, Tolerability and Immunogenicity of INO-4800, a Prophylactic Vaccine Against SARS-CoV-2, Administered Intradermally Followed by Electroporation in Healthy Volunteers
Brief Title: Safety, Tolerability and Immunogenicity of INO-4800 for COVID-19 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: COVID19-001
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus Infection
Keywords: DNA vaccine; Electroporation
MeSH Terms: conditions — Coronavirus Infections | interventions — reluscovtogene ralaplasmid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Group 1: INO-4800 (Experimental): Participants will receive one ID injection of 1.0 milligram (mg) of INO-4800 followed by EP using the CELLECTRA® 2000 device per dosing visit.
  Interventions: Drug: INO-4800; Device: CELLECTRA® 2000
- Group 2: INO-4800 (Experimental): Participants will receive two ID injections of 1.0 mg (total 2.0 mg per dosing visit) of INO-4800 followed by EP using the CELLECTRA® 2000 device per dosing visit.
  Interventions: Drug: INO-4800; Device: CELLECTRA® 2000
- Group 3: INO-4800 (Experimental): Participants will receive one ID injection of 0.5 mg of INO-4800 followed by EP using the CELLECTRA® 2000 device per dosing visit.
  Interventions: Drug: INO-4800; Device: CELLECTRA® 2000

INTERVENTIONS:
Drug: INO-4800 — INO-4800 will be administered ID on Day 0, Week 4 and at the optional Booster Dose Visit.
Device: CELLECTRA® 2000 — EP using the CELLECTRA® 2000 device will be administered following ID delivery of INO-4800 on Day 0, Week 4 and at the optional Booster Dose Visit.

SUMMARY:
This is an open-label trial to evaluate the safety, tolerability and immunological profile of INO-4800 administered by intradermal (ID) injection followed by electroporation (EP) using CELLECTRA® 2000 device in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Judged to be healthy by the Investigator on the basis of medical history, physical examination and vital signs performed at screening.
* Able and willing to comply with all study procedures.
* Screening laboratory results within normal limits or deemed not clinically significant by the Investigator.
* Body Mass Index of 18-30 kg/m^2, inclusive, at screening.
* Negative serological tests for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody and Human Immunodeficiency Virus (HIV) antibody at screening.
* Screening electrocardiogram (ECG) deemed by the Investigator as having no clinically significant findings (e.g. Wolff-Parkinson-White syndrome).
* Use of medically effective contraception with a failure rate of < 1% per year when used consistently and correctly from screening until 3 months following last dose, be post-menopausal, be surgically sterile or have a partner who is sterile.

Exclusion Criteria:

* Pregnant or breastfeeding or intending to become pregnant or father children within the projected duration of the trial from screening until 3 months following last dose.
* Is currently participating in or has participated in a study with an investigational product within 30 days preceding Day 0.
* Previous exposure to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or receipt of an investigational product for the prevention or treatment of COVID-19, middle east respiratory syndrome (MERS), or severe acute respiratory syndrome (SARS).
* In a current occupation with high risk of exposure to SARS-CoV-2 (e.g., health care workers or emergency response personnel having direct interactions with or providing direct care to patients).
* Current or history of the following medical conditions:

  * Respiratory diseases
  * Hypersensitivity or severe allergic reactions to vaccines or drugs
  * Diagnosis of diabetes mellitus
  * Hypertension
  * Malignancy within 5 years of screening
  * Cardiovascular diseases
* Immunosuppression as a result of underlying illness or treatment including:

  * Primary immunodeficiencies
  * Long term use (≥7 days) of oral or parenteral glucocorticoids
  * Current or anticipated use of disease-modifying doses of anti-rheumatic drugs and biologic disease-modifying drugs
  * History of solid organ or bone marrow transplantation
  * Prior history of other clinically significant immunosuppressive or clinically diagnosed autoimmune disease
* Fewer than two acceptable sites available for intradermal (ID) injection and electroporation (EP) considering the deltoid and anterolateral quadriceps muscles.
* Reported smoking, vaping, or active drug, alcohol or substance abuse or dependence.
* Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Baseline up to Week 52 (if not receiving an optional booster dose) or the 48 Week Post-Booster Dose Visit (if receiving an optional booster dose)
Percentage of Participants with Administration (Injection) Site Reactions | Day 0 up to Week 52 (if not receiving an optional booster dose) or the 48 Week Post-Booster Dose Visit (if receiving an optional booster dose)
Percentage of Participants with Adverse Events of Special Interest (AESIs) | Baseline up to Week 52 (if not receiving an optional booster dose) or the 48 Week Post-Booster Dose Visit (if receiving an optional booster dose)
Change from Baseline in SARS-CoV-2 Spike Glycoprotein Antigen-Specific Binding Antibody Titers | Baseline up to Week 52 (if not receiving an optional booster dose) or the 48 Week Post-Booster Dose Visit (if receiving an optional booster dose)
Change from Baseline in Antigen-Specific Cellular Immune Response | Baseline up to Week 52 (if not receiving an optional booster dose) or the 48 Week Post-Booster Dose Visit (if receiving an optional booster dose)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ning Jiang, MD PhD, Study Director — Inovio Pharmaceuticals
Locations (3):
- United States (3):
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and all collected IPD will be stripped of identifiers and may be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Anonymous IPD may be shared following or during the publication of summary data. Archival data may be accessed for up to 10 years following the end of the study.
Access Criteria: Those who request the anonymous IPD must provide a plan of study explaining how the data will be used. Requests may be sent to the Central Contact Person. Requests will be reviewed based on the potential for the planned use of the IPD for advancing scientific knowledge and theory.

REFERENCES:
- [Derived] Kraynyak KA, Blackwood E, Agnes J, Tebas P, Giffear M, Amante D, Reuschel EL, Purwar M, Christensen-Quick A, Liu N, Andrade VM, Diehl MC, Wani S, Lupicka M, Sylvester A, Morrow MP, Pezzoli P, McMullan T, Kulkarni AJ, Zaidi FI, Frase D, Liaw K, Smith TRF, Ramos SJ, Ervin J, Adams M, Lee J, Dallas M, Shah Brown A, Shea JE, Kim JJ, Weiner DB, Broderick KE, Humeau LM, Boyer JD, Mammen MP. SARS-CoV-2 DNA Vaccine INO-4800 Induces Durable Immune Responses Capable of Being Boosted in a Phase 1 Open-Label Trial. J Infect Dis. 2022 Jun 1;225(11):1923-1932. doi: 10.1093/infdis/jiac016. PMID 35079784
- [Derived] Tebas P, Yang S, Boyer JD, Reuschel EL, Patel A, Christensen-Quick A, Andrade VM, Morrow MP, Kraynyak K, Agnes J, Purwar M, Sylvester A, Pawlicki J, Gillespie E, Maricic I, Zaidi FI, Kim KY, Dia Y, Frase D, Pezzoli P, Schultheis K, Smith TRF, Ramos SJ, McMullan T, Buttigieg K, Carroll MW, Ervin J, Diehl MC, Blackwood E, Mammen MP, Lee J, Dallas MJ, Brown AS, Shea JE, Kim JJ, Weiner DB, Broderick KE, Humeau LM. Safety and immunogenicity of INO-4800 DNA vaccine against SARS-CoV-2: A preliminary report of an open-label, Phase 1 clinical trial. EClinicalMedicine. 2021 Jan;31:100689. doi: 10.1016/j.eclinm.2020.100689. Epub 2020 Dec 24. PMID 33392485